CLINICAL TRIAL: NCT04632394
Title: Can MRI-based Computational Modelling of the Heart be Used to Predict Critical Substrate in Scar-dependent Ventricular Tachycardia Ablation?
Brief Title: Multimodality Assessment of Ventricular Scar Arrhythmogenicity.
Status: Completed | Type: Observational
Sponsor: St George's, University of London (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020.0237
Record Dates: First submitted 2020-10-20; First posted 2020-11-17 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2023-04

CONDITIONS: Ventricular Tachycardia
Keywords: ventricular tachycardia; ablation; cardiac MRI; computational modelling
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Patients with scar-dependent ventricular tachycardia, requiring ablation. These patients will have satisfied the inclusion/exclusion criteria and be put forward for VT ablation. They will undergo the previously described study protocol, including generation of a computational model of the heart from their cardiac MRI and a VT ablation where we will study the points of interest generated from the MRI model in detail.
  Interventions: Diagnostic Test: Generation of computational model from cardiac MRI.; Procedure: VT ablation

INTERVENTIONS:
Diagnostic Test: Generation of computational model from cardiac MRI. — Routine cardiac MRI scan results will be sent to Johns Hopkins University where a computer-generated model of the heart will be made, which will demonstrate predicted areas critical to VT generation and maintenance. This data will be sent back to St George's, and integrated with the standard VT ablation mapping software to allow comparison of its accuracy with standard mapping techniques.
Procedure: VT ablation — Routine VT ablation as described elsewhere in the literature. However, a brief period of extra time (~30 minutes) will be spent analysing the areas of the heart which the MRI scan predicted as being important for generation of VT. We will study the effect of ablation of these areas (if indicated) on distant parts of the heart.

SUMMARY:
We aim to improve our understanding of a life-threatening heart rhythm disorder known as ventricular tachycardia (VT). This is a disorder which originates from the lower chamber of the heart and frequently is associated with heart disease. We will use an MRI scan to generate a computer based model of the heart which can predict areas of the heart which are important in generating this rhythm disorder. We intend to assess how accurate this computer model is compared to traditional invasive assessment of the heart muscle. We also aim to assess the electrical characteristics of those areas which were predicted by the computer model in order to see why they were thought to be so important.

All patients seen at St George's Hospital with VT will be eligible. As is routine for these patients, they will have an MRI scan of the heart. We will then use this scan to create a virtual reconstruction of the heart from which predictions of the critical areas of the heart which are generating the rhythm problem will be made. Then we will perform a VT ablation (studying the electrical properties and if necessary making a burn to treat the rhythm problem) - as per standard of care, however during the ablation we will spend extra time collecting information comparing the accuracy of the computer-generated model to the traditional invasive signals which guide ablation. We will study the electrical properties of those predicted areas to see what is special about them. The study will last up to three years.

DETAILED DESCRIPTION:
Patients will be eligible for this trial both from referrals as an outpatient, where VT has been detected on a heart rhythm monitor or ECG (electrical heart tracing), or as an inpatient where they have been admitted to hospital with symptoms of VT. Our study investigators will discuss the research with the patient and give them the relevant information in an understandable format as part of a Patient Information Sheet so that they can make an informed decision about whether or not to participate in the research.

An MRI scan of the heart is a standard investigation for patients presenting with VT, however if the patient is included in the study, the MRI scan images will be anonymised and sent confidentially to the Institute of Computational Modelling at Johns Hopkins University in USA where the images will be reconstructed into a 3D representation of the patients heart, where the electrical pathways and source of the VT can be seen. This information will be sent back (again confidentially and anonymously) to St George's Hospital in time for their routine VT ablation procedure.

During the VT ablation The MRI scan model will be combined with the invasively-obtained information and we will assess the various areas of the heart which are responsible for the VT, particularly relating to areas of scar within the heart, which are frequently seen in these patients. We will assess the electrical properties of the areas highlighted as the cause of the VT from the MRI scan.

We will assess the accuracy of the computer model compared to the traditional invasive measurements that we take. We will first ablate those areas of the heart which the model predicted as being important (as long as the invasive characteristics support ablation there) and then see what effect this had on the electrical properties of other areas of the heart. However, we will not ablate any area of the heart based solely on the MRI model; it will only influence the order of ablation and not tell us whether to ablate or not.

The procedure can take 4-6 hours in total. The extra information gathered as part of the research protocol may extend this by a maximum of 10%. No extra pieces of equipment, procedures or medications are involved in the research, just the time taken to generate a computer model of the heart as well as a extra time to assess the heart in more detail during the ablation.

Following the ablation, the patients will be followed at 3, 6 and 12 months with a heart rhythm monitor and a clinical review as an outpatient as per routine standard of care. From this, we will collect data on frequency of recurrence of rhythm disturbance, therapy from their implantable cardioverter-defibrillators, symptoms and complications following the ablation procedure.

The information gathered during the procedure will be analysed and research papers generated from the results.

ELIGIBILITY:
Inclusion Criteria:

Adult inpatients admitted to St George's Hospital London with sustained ventricular tachycardia or outpatients identified from the arrhythmia clinic with significant monomorphic ventricular tachycardia noted on cardiac monitoring who:

* Have sustained, monomorphic scar-dependent ventricular tachycardia
* Are symptomatic
* Failed, unable or unwilling to tolerate anti-arrhythmic medications
* Able to have a cardiac MRI
* Have a life expectancy > 1 year
* At least 40 days following a myocardial infarction

Exclusion Criteria:

* Patients under the age of 18
* Patients who are unable to give informed consent
* Pregnant patients
* Unable to have cardiac MRI
* Prohibitive procedural risk
* Unable to tolerate the ablation procedure due to haemodynamic instability

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study setting is a large tertiary centre hospital in London, St George's University Hospital which serves a population of around 1.3 million. It also receives referrals from district general hospitals in the surrounding area. Referrals are made to a specialist arrhythmia clinic from which suitable patients can be identified. The majority of recruited patients are expected to be outpatients who are symptomatic from VT despite optimal medical therapy. This will allow sufficient time to perform the cardiac MRI and to generate the computational model. In some scenarios, emergency admissions with symptomatic VT may be included if they are suitable for inpatient VT ablation and there is sufficient time for the MRI and computation analysis to take place prior to the VT ablation.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-04-02 (Actual); Study Completion 2024-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Magdi Saba, MD, Study Director — St George's Hospital / SGUL; Anthony Li, MD, Study Director — St George's Hospital
Locations (1):
- St George's University Hospitals NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Not applicable - participant data will not be shared with other researchers outside the study group.

REFERENCES:
- [Derived] Waight MC, Prakosa A, Li AC, Bunce N, Marciniak A, Trayanova NA, Saba MM. Personalized Heart Digital Twins Detect Substrate Abnormalities in Scar-Dependent Ventricular Tachycardia. Circulation. 2025 Feb 25;151(8):521-533. doi: 10.1161/CIRCULATIONAHA.124.070526. Epub 2025 Jan 6. PMID 39758009

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cases
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort: Cohort of patients who underwent digital twin generation and VT ablation.
Arm/Group | Cohort
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 14
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 18

OUTCOME MEASURES:

1. Primary Outcome: Electrogram Duration at Digital Twin Predicted Sites Compared to Non-predicted Sites
Description: Duration of electrograms at digital twin predicted sites compared to non-predicted sites on invasive mapping within areas of bipolar low voltage (<1.5mV)
Time Frame: During ablation
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Predicted Sites: Digital twin sites predicted to harbour VT
- Non-predicted Sites: Sites not suggestive of critical importance by the digital twin
Arm/Group | Predicted Sites | Non-predicted Sites
Number analyzed (Participants) | 18 | 18
ms | 77.5 (25.8) | 65.7 (40.0)

2. Secondary Outcome: Symptom Assessment at 12 Month Clinical Follow up
Description: Assessment of patient's symptoms at a clinical consultation following the ablation.
Time Frame: 12 months
Population: Recurrence of ventricular arrhythmia at 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Cases
Number analyzed (Participants) | 18
Participants | 2

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Cases
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 1/18
Other Adverse Events (participants affected / at risk) | 0/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cases (N=18)
Ventricular septal defect (Cardiac disorders) | 1 (1) — Late presenting VSD in one patient with NICM following ablation to the basal septum which was thinned pre-ablation. Managed conservatively.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04632394/Prot_SAP_000.pdf
  • Informed Consent Form (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/94/NCT04632394/ICF_001.pdf